CLINICAL TRIAL: NCT05618496
Title: Multi-centre, Open-label, First-in-man Study With Epipad Used in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contipro Pharma a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-EPI-1_09-20
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with Epipad (Experimental): Epipad
  Interventions: Device: Sodium Hyaluronate Lyophilizate

INTERVENTIONS:
Device: Sodium Hyaluronate Lyophilizate — Device is placed directly onto the treated wound. The wound should be cleaned with antiseptic solution prior to the device administration. The device is fixed on the wound by secondary dressing: e.g. plaster, compression.
  Other Names: Epipad

SUMMARY:
The main objective of the trial is to confirm safety of a new product - Epipad. The main impact of the device is to provide good environment for the healing of chronic wounds and wounds in the last healing phase (granulation and epithelisation).

ELIGIBILITY:
Inclusion Criteria:

* Patient suffered from superficial wound of different etiology
* Wounds in terminal phase of healing
* Wounds without visible sign of infection
* Max. size of the wound: 10 x 20 cm (i.e. two pieces of the product)
* Duration of wound treatment of at least 6 weeks
* Subject willing and able to provide written informed consent
* Ability to communicate well with the investigator in local language, and to understand and comply with the requirements of the study

Exclusion Criteria:

* Sloughy or necrotic wound bed
* Severely contaminated or infected wound
* Age < 18 years
* Pregnant or lactating woman
* Subject in terminal stage of living
* Subject with cancer disease
* Subject with known hypersensitivity or allergy to any component of the investigational device
* Subject participating in other interventional clinical trial
* Alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in the wound dimensions (width x length) | Week 3
  Change in the wound dimensions from baseline

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - Fakultni nemocnice u sv. Anny, Brno
  - Levitovo centrum nasledne pece, Hořice
  - Vojenska nemocnice Olomouc, Olomouc
  - Vsetinska nemocnice, Vsetín

IPD SHARING:
Plan to Share IPD: No